CLINICAL TRIAL: NCT04964726
Title: Dyadic Neurofeedback for Emotion Regulation in Youth With Maternal Adversity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHS2021035
Record Dates: First submitted 2021-06-25; First posted 2021-07-16 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Emotional Dysfunction; Early Life Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real-time fMRI dyadic neurofeedback (Experimental)
  Interventions: Behavioral: Real-time fMRI dyadic neurofeedback

INTERVENTIONS:
Behavioral: Real-time fMRI dyadic neurofeedback — Participants will attempt to regulate their partner's brain activation in a specified brain region via real-time fMRI neurofeedback.

SUMMARY:
This study will examine the effect of a real-time functional magnetic resonance imaging (fMRI) dyadic neurofeedback protocol with mothers and their adolescent daughters. Mothers will view a moving bar showing their daughters' brain activity on a computer screen while talking to their daughters.

DETAILED DESCRIPTION:
The current study will determine the effects of a real-time functional magnetic resonance imaging dyadic neurofeedback (rtfMRI-DNF) protocol that will train mothers with a history of adverse childhood experiences (ACEs) to regulate adolescents' activation in the anterior insular cortex (aIC) - a key brain region for ER. The proposed study will test the efficacy of this protocol to promote healthy ER-related neurodevelopment in adolescents with a maternal history of adversity. The proposed study will use DNF to provide neurofeedback from the adolescent's aIC to the parent as the parent and adolescent engage in an emotion discussion task together. Parents and adolescents (n=10 dyads) will communicate via microphones and noise-canceling headphones while the adolescent is undergoing fMRI scanning. Specific aims of the current study are: (1) to determine the brain response to aIC DNF adolescents, and (2) to determine effects of DNF on parenting behaviors. This study is significant because engaging with parents in DNF can promote positive ER development in adolescents at risk due to the intergenerational effects of ACEs.

ELIGIBILITY:
Inclusion Criteria:

All participants inclusion criteria:

* Biological female
* Sufficient English fluency to complete tasks
* Co-residing at least 4 days per week

Inclusion criteria for adult participants:

* Primary caregiver for more than 50% of child's lifespan
* History of at least two adverse childhood experiences
* Biological parent of adolescent participant

Inclusion criteria for adolescents:

* Eligible for fMRI
* Right-handed
* Body mass index between 16 and 40 (inclusive)
* Age 14-17 years

Exclusion Criteria:

Exclusion criteria for all participants:

* Current psychiatric diagnosis

Exclusion criteria for adolescent participants:

* Neurodevelopmental delay
* History of psychiatric disorder
* Medications influencing fMRI
* Medical conditions influencing fMRI

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Parent report of child's gender identity as "girl"
Enrollment: 30 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level-Dependent (BOLD) signal changes (brain activation) | One hour (measured during first scan session)
  Activation in the brain region targeted for neurofeedback and associated regions at Session 1. We hypothesize that lower activity will indicate a better outcome.
Blood Oxygen Level-Dependent (BOLD) signal changes (brain activation) | One hour (measured during second scan session)
  Activation in the brain region targeted for neurofeedback and associated regions at Session 2. We hypothesize that lower activity will indicate a better outcome.
Resting-state network activity (change over time) | Change in resting-state activity over one week, from Session 1 to Session 2. Resting-state scan will last approximately 8 minutes.
  Brain activity during fMRI resting-state scan
Parent validating statements (change over time) | Change in frequency in validation as coded by the manual over one week, from Session 1 to Session 2. Validating statements are measured and recorded during the scan sessions.
  Validating statements made by the parent participant during the scan sessions. Statements will be coded using the Parent-Child Validation/Invalidation Behavior Coding Scales (Schneider & Fruzzetti, 2002). Higher scores are indicative of a better outcome.

SECONDARY OUTCOMES:
Parenting behaviors (change over time) | Measured at the first research session and biweekly for two months
  Change over time in adolescent's responses to the Children's Report of Parent Behavior Inventory (Schludermann & Schludermann, 1988). The CRPBI has 3 subscales, each with a score range of 10-30. Interpretation/valence of the scores varies by subscale.
Emotion regulation (change over time) | Measured at the first research session and biweekly for two months
  Change over time in adolescent's responses to the Difficulties in Emotion Regulation Scale (Gratz & Roemer, 2008). The DERS consists of 36 items rated on a 1-5 Likert scale (scale range: 36-180). Higher scores indicate greater difficulties with emotion regulation.
Depressive symptoms (change over time) | Measured at the first research session and biweekly for two months
  Change over time in adolescent's responses to the PROMIS (Patient Reported Outcome Measurement Information System) Pediatric Short Form Version 2 (Quinn et al., 2014). This is an 8-item scale with scores ranging from 8-40, with higher scores indicating more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hardesty Center for Clinical Research and Neuroscience, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes